CLINICAL TRIAL: NCT00958984
Title: Continuous Hemoglobin and Plethysmograph Variability Index Monitoring May Provide Superior Assessment During Visceral Solid Organ Transplantation in Children: a Prospective Cohort Study
Brief Title: Continuous Hemoglobin Monitoring in Pediatric Transplant
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Other Study IDs: 0294-09-FB
Record Dates: First submitted 2009-08-13; First posted 2009-08-14 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Pediatric Solid Organ Transplant
Keywords: pediatric; solid organ transplant; hemoglobin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine the clinical utility of non-invasive monitoring of Hemoglobin (Hgb) and Plethysmograph Variability Index (PVI) values during the intraoperative period of visceral solid organ transplantation in children. Hemoglobin values reflect oxygen-carrying capacity of the blood and PVI reflects fluid balance and perfusion.

DETAILED DESCRIPTION:
Background and Significance: The pediatric visceral solid organ transplant patient experiences significant hemodynamic changes and anemia during the process of transplantation. These changes occur as a result of several factors: 1) Concomitant high output cardiac failure found with liver failure causes an increased sensitivity to modest decreases in intravascular volume resulting in hypotension and shock; 2) Patients may experience significant blood loss [2 to 6 times circulating blood volume] during the operative period; 3) Replenishment of intravascular volume based on intermittent hgb measurements, estimates of blood loss and hemodynamic insufficiency leads to prolongation of anemia and/or development of polycythemia. Continuous monitoring of hgb and PVI should prove superior to current procedure to determine intravascular volume depletion, anemia and prevent polycythemia. Based on the findings of this study, an intraoperative treatment algorithm can be developed for the efficacious and judicious use of blood products and fluids during resuscitation and improved perioperative management of the pediatric transplant patient.

Specific Aims: 1) Determine the severity, time of onset, and duration of PVI variability consistent with hypovolemia in relation to organ explantation, vascular clamping, reperfusion of newly transplanted organ(s) and bleeding events. 2) Determine the severity, time of onset, and duration of anemia (hgb < 8 gm/dL) and polycythemia (hgb > 13 gm/dL) in relation to these events. 3) Determine if the administration of blood products, crystalloid, and colloid solutions based on subjective assessment of hemodynamic indices, blood loss and intermittent hemoglobin measurement leads to inappropriate intraoperative resuscitation .

Preliminary Data: Episodic hemoglobin sampling during transplantation in 13 pediatric patients at NMC revealed the following: anemic values occurred in 69% (9/13) of the patients, with 38% (5/13) of those having 3 or more anemic values (lowest hgb: 1.7g/dL); polycythemic values occurred in 13% (2/13) of the patients (highest hgb: 14.8g/ dL). All patients displayed hypotension during the operative period despite having CVP measurements that matched pre-transplant values. During a recent introductory session for the Masimo Rainbow SET monitor and sensor probe, a toddler undergoing liver, small bowel, and pancreas transplant was observed and hemoglobin values were noted from both the Masimo monitor and conventional episodic blood sampling. Values obtained from both sources simultaneously revealed ≤ 1 g/dL discrepancy between the measurement methods in 100% of the values.

Research Protocol: Twenty-one subjects ≤18 years of age undergoing solid organ transplant, will be monitored during the intraoperative period transcutaneously for continuous PVI and hgb. Data collection will also include continuous CVP and MAP, significant operative events, concurrent blood loss, fluid administration, and conventional episodic Hgb sampling. Data from the hospital monitoring system will be time synchronized with Masimo derived measurements. The research team will coordinate recording of all events in the intra-operative period using standardized case report forms. Anesthesiologist and transplant team are blinded to Masimo data. Continuous Hgb and PVI will not be used to determine clinical treatment. The expected duration of this study will be two years based on the average number of pediatric solid organ transplant procedures participated in by the Anesthesiology Department at The Nebraska Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* age between birth up to, and including, 18 years
* undergoing solid organ transplantation at The Nebraska Medical Center
* signed informed consent and assent as applicable

Exclusion Criteria:

* prospective subjects already under the effects of anesthesia

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients under age 19 years of age undergoing visceral solid organ transplant at The Nebraska Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2009-08-11 (Actual); Primary Completion 2011-08-01 (Actual); Study Completion 2011-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Sullivan, MD, Principal Investigator — University of Nebraska
Locations (1):
- Unversity of Nebraska Medical Center, Omaha, Nebraska, United States